CLINICAL TRIAL: NCT05765682
Title: Mepivacaine Vs. Bupivacaine Spinal: Effect on Return of Motor Function, Time to Ambulation, and Length of Stay in Total Knee Arthroplasty
Brief Title: Mepivacaine Vs. Bupivacaine Spinal for TKA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Clinton F. Pillow, Physician, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Pro00125382
Record Dates: First submitted 2023-01-27; First posted 2023-03-13 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Total Knee Replacement

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Subject, surgeon, and care team members will be blinded to the assigned randomization group. The anesthesiologist will not be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mepivacaine Spinal (Active Comparator): Mepivacaine (60 mg: 3ml of 2%) or will be injected into the intrathecal space.
  Interventions: Other: Mepivacaine Spinal
- Bupivacaine Spinal (Active Comparator): Isobaric bupivacaine (10mg: 2ml or 0.5%) will be injected into the intrathecal space.
  Interventions: Other: Bupivacaine Spinal

INTERVENTIONS:
Other: Mepivacaine Spinal — spinal block using 60mg of mepivacaine
  Arms: Mepivacaine Spinal
Other: Bupivacaine Spinal — spinal block using 10mg of bupivacaine
  Arms: Bupivacaine Spinal

SUMMARY:
This study will enroll patients 18-75 years of age who are undergoing elective primary total knee replacement. The patients will be randomized to receive one of two spinal blocks: 1) mepivacaine or 2) bupivacaine. The primary goal is to determine which group arrives at recovery of motor function first. Ultimately, this study will explore if mepivacaine leads to earlier return of motor function and ultimately earlier movement and discharge times following total knee replacement.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-75 years of age
* Undergoing elective primary total knee arthroplasty

Exclusion Criteria:

* Inability to ambulate or impaired motor function in lower extremities prior to surgery
* Contraindication to spinal anesthetic
* Taking over 30mg oxycodone per day (or calculated MME equivalent)
* Subjects that are unable or choose not to give informed consent
* Known preoperative substance abuse
* Pregnant women
* Allergy to all opioids

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2023-03-13 (Actual); Primary Completion 2024-08-23 (Actual); Study Completion 2024-08-25 (Actual)

PRIMARY OUTCOMES:
Time until return of motor function following spinal placement | From anesthesia stop time until 7 days post-op
  This will be defined as full strength with both 1) foot plantar and dorsiflexion and 2) hip flexion and 3) knee flexion in the non-operative extremity.

SECONDARY OUTCOMES:
Ambulation | from anesthesia stop time until 7 days post-op
  Time to first ambulation and distance at first ambulation
Length of Stay | Time from anesthesia end time to when discharge order is written, up to 30 days post-op
  based on anesthesia end time to time discharge order written
Side Effects | 0-48 hours post spinal placement
  Side effects such as Urinary retention, dizziness, symptomatic hypotension, transient neurologic symptoms
Pain Scores | Pacu to 48 hours post-spinal placement
  Visual Analog Pain Score 0-100 pain scores at rest, and with movement. A lower pain score means a better outcome.

OTHER OUTCOMES:
Preoperative opioid use | within past 90 days at time of procedure
  Use of opioids in the pre-operative period converted to MME (morphine equivalent)
Tourniquet use | during procedure for up to 7 days hours after procedure ends
  Whether or not a tourniquet is used during surgery will be recorded as yes or no.
Cement use | during procedure or up to 7 days hours after procedure ends
  Whether or not a cement is used during surgery will be recorded as yes or no.
Robotic or not | during procedure or up to 7 days hours after procedure ends
  Whether or not the procedure is robotic or not will be recorded as yes or no.

CONTACTS AND LOCATIONS:
Overall Officials: Clinton Pillow, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pillow CF, Brewbaker C, Wolf BJ, Barrett W, Hansen E, Brown A, Crawford D, Wilson SH. Mepivacaine versus bupivacaine spinal anesthesia for return of motor function following total knee arthroplasty: a randomized controlled trial. Reg Anesth Pain Med. 2025 May 1:rapm-2024-106342. doi: 10.1136/rapm-2024-106342. Online ahead of print. PMID 40316299